CLINICAL TRIAL: NCT06655675
Title: Changes in Velocimetric Indices of Uterine and Umbilical Arteries Before and After Combined Spinal-epidural Analgesia in Laboring Women (PART I and PART II)
Brief Title: Changes in Velocimetric Indices of Uterine and Umbilical Arteries Before and After Combined Spinal-epidural Analgesia in Laboring Women (PART II)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 24-09
Record Dates: First submitted 2024-10-17; First posted 2024-10-23 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Labor Pain
Keywords: combined spinal epidural (CSE); fetal bradycardia; ultrasound; velocimetric index; hypertension
MeSH Terms: conditions — Labor Pain; Hypertension | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ultrasound - patients without hypertensive disorders of pregnancy (Experimental): Ultrasound will be used to measure velocimetric index of the umbilical artery.
  Interventions: Device: Ultrasound
- Ultrasound - patients with diagnosed hypertensive disorders of pregnancy (Experimental): Ultrasound will be used to measure velocimetric index of the umbilical artery.
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: Ultrasound — Ultrasound scan of the umbilical artery

SUMMARY:
Combined spinal-epidural (CSE) for labor analgesia has been used for many years and is practiced commonly at our institution, especially when the patient requests immediate pain relief. CSE is not only beneficial for its faster onset of analgesia, but also it is favorable in relation to the need for rescue analgesia, urinary retention, and rate of instrumental delivery compared to the traditional epidural. Despite its beneficial effects, there is a risk of about 15-30% of developing abnormal fetal heart rate following CSE. This is self-resolving with minimal or no intervention. Although the cause of fetal bradycardia is not fully elucidated, variations in uterine artery blood flow after epidural analgesia are thought to be due to the interaction of numerous events related to blockade of sympathetic innervations, fluid administration, maternal hypotension, uterine vascular effects of sympathetic block, fluctuations in circulating catecholamines, and possibly the effect of opioids. Similar mechanism is thought to be a cause of fetal bradycardia after the CSE with its faster onset and superior block.

Maternal or fetal circulation during labor can be assessed using continuous-wave Doppler ultrasound to monitor maternal uterine artery (UtA) and fetal umbilical artery (UmA) velocity waveforms to detect changes in blood flow. The velocimetry indices mentioned above have been often used to assess the changes in the blood flow before and after the induction of epidural analgesia during labor in several studies. Although there are some studies regarding the effect of labor epidural analgesia using velocimetry indices, but there is currently no published study evaluating velocimetry indices of uterine and umbilical arteries before and after the induction of CSE. Thus, the aim of this study is to investigate the impact of CSE to maternal and fetal blood flow to evaluate the relationships.

The investigators hypothesize that both uterine artery and umbilical artery blood flow are reduced after the induction of CSE, which may be responsible for the occurrence of fetal bradycardia.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Term pregnant patients requesting labor analgesia
* Singleton pregnancy
* Term pregnant patients in active labor
* ASA<4
* No evidence of fetal congenital anomalies, fetal compromise or fetal decelerations prior to CSE
* Patients with and without diagnosed hypertensive disorders of pregnancy

Exclusion Criteria:

* Refusal to consent for the study
* Known spinal deformities
* Previous back instrumentation
* Patients with BMI>50 kg/㎡ due to anticipated technical challenges in Doppler studies

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-10-30 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Umbilical artery velocimetric index - systolic/diastolic ratio (S/D) at 10 minutes | 10 minutes
  Umbilical artery velocimetric index - systolic/diastolic ratio (S/D) will be measured 10 minutes after combined spinal epidural, with the uterus in relaxed and contracted states.
Umbilical artery velocimetric index - pulsatility index (PI) at 10 minutes | 10 minutes
  Umbilical artery velocimetric index - pulsatility index (PI) will be measured 10 minutes after combined spinal epidural, with the uterus in relaxed and contracted states.
Umbilical artery velocimetric index - resistance index (RI) at 10 minutes | 10 minutes
  Umbilical artery velocimetric index - resistance index (RI) will be measured 10 minutes after combined spinal epidural, with the uterus in relaxed and contracted states.

SECONDARY OUTCOMES:
Umbilical artery velocimetric index - systolic/diastolic ratio (S/D) at baseline | 5 minutes
  Umbilical artery velocimetric index - systolic/diastolic ratio (S/D) will be measured prior to combined spinal epidural, with the uterus in relaxed and contracted states.
Umbilical artery velocimetric index - pulsatility index (PI) at baseline | 5 minutes
  Umbilical artery velocimetric index - pulsatility index (PI) will be measured prior to combined spinal epidural, with the uterus in relaxed and contracted states.
Umbilical artery velocimetric index - resistance index (RI) at baseline | 5 minutes
  Umbilical artery velocimetric index - resistance index (RI) will be measured prior to combined spinal epidural, with the uterus in relaxed and contracted states.
Umbilical artery velocimetric index - systolic/diastolic ratio (S/D) at 5 minutes | 5 minutes
  Umbilical artery velocimetric index - systolic/diastolic ratio (S/D) will be measured 5 minutes after combined spinal epidural, with the uterus in relaxed and contracted states.
Umbilical artery velocimetric index - pulsatility index (PI) at 5 minutes | 5 minutes
  Umbilical artery velocimetric index - pulsatility index (PI)will be measured 5 minutes after combined spinal epidural, with the uterus in relaxed and contracted states.
Umbilical artery velocimetric index - resistance index (RI) at 5 minutes | 5 minutes
  Umbilical artery velocimetric index - resistance index (RI) will be measured 5 minutes after combined spinal epidural, with the uterus in relaxed and contracted states.
Umbilical artery velocimetric index - systolic/diastolic ratio (S/D) at 20 minutes | 20 minutes
  Umbilical artery velocimetric index - systolic/diastolic ratio (S/D) will be measured 20 minutes after combined spinal epidural, with the uterus in relaxed and contracted states.
Umbilical artery velocimetric index - pulsatility index (PI) at 20 minutes | 20 minutes
  Umbilical artery velocimetric index - pulsatility index (PI) will be measured 20 minutes after combined spinal epidural, with the uterus in relaxed and contracted states.
Umbilical artery velocimetric index - resistance index (RI) at 20 minutes | 20 minutes
  Umbilical artery velocimetric index - resistance index (RI) will be measured 20 minutes after combined spinal epidural, with the uterus in relaxed and contracted states.
Umbilical artery velocimetric index - systolic/diastolic ratio (S/D) at 30 minutes | 5 minutes
  Umbilical artery velocimetric index - systolic/diastolic ratio (S/D) will be measured 30 minutes after combined spinal epidural, with the uterus in relaxed and contracted states.
Umbilical artery velocimetric index - pulsatility index (PI) at 30 minutes | 30 minutes
  Umbilical artery velocimetric index - pulsatility index (PI) will be measured 30 minutes after combined spinal epidural, with the uterus in relaxed and contracted states.
Umbilical artery velocimetric index - resistance index (RI) at 30 minutes | 30 minutes
  Umbilical artery velocimetric index - resistance index (RI) will be measured 30 minutes after combined spinal epidural, with the uterus in relaxed and contracted states.
Pain score at baseline - questionnaire | 1 minute
  Pain score - verbal numeric rating scale (0-10) prior to combined spinal epidural
Pain score at 10 minutes - questionnaire | 10 minutes
  Pain score - verbal numeric rating scale (0-10) at 10 minute after combined spinal epidural
Pain score at 30 minutes - questionnaire | 30 minutes
  Pain score - verbal numeric rating scale (0-10) at 30 minute3 after combined spinal epidural
Sensory block level at 10 minutes | 10 minutes
  Sensory block level at 10 minutes following combined spinal epidural
Sensory block level at 30 minutes | 30 minutes
  Sensory block level at 30 minutes following combined spinal epidural
frequency of uterine contractions | 10 minutes
  The number of contractions on the monitor in a 10 minute period.
Presence of prolonged hypertonic uterine contractions- questionnaire | 30 minutes
  Presence of prolonged hypertonic uterine contractions as measured by the monitor
Hypotension: systolic blood pressure less than 80% of baseline | 30 minutes
  Systolic blood pressure < 80% of baseline, monitored q5 for 30 minutes following combined spinal epidural
Hypertension: systolic blood pressure greater than 120% of baseline | 30 minutes
  Systolic blood pressure > 120% of baseline, monitored q5 for 30 minutes following combined spinal epidural
Bradycardia: heart rate less than 70% of baseline | 30 minutes
  Heart rate < 70% of baseline or a heart rate < 50bpm, monitored q5 for 30 minutes following combined spinal epidural
Desaturation: oxygen level <95% | 30 minutes
  Oxygen level <95%, monitored q5 for 30 minutes following combined spinal epidural
fetal heart rate at baseline | 5 minutes
  fetal heart rate at baseline, prior to combined spinal epidural
fetal heart rate q5 min up to 30 minutes | 30 minutes
  fetal heart rate q5 min up to 30 minutes following combined spinal epidural
presence of fetal bradycardia - questionnaire | 30 minutes
  presence of fetal bradycardia (fetal heart rate <110)
presence of fetal prolonged deceleration - questionnaire | 30 minutes
  presence of fetal prolonged deceleration (fetal heart rate <110/min lasting less than 10 minutes)
presence of fetal persistent late decelerations - questionnaire | 30 minutes
  presence of fetal persistent late decelerations will be recorded
presence of fetal non-reassuring variable deceleration - questionnaire | 30 minutes
  presence of fetal non-reassuring variable deceleration will be recorded
presence of fetal salutatory variability - questionnaire | 30 minutes
  presence of fetal salutatory variability (FHR change>25beats) will be recorded
Neonatal weight | up to 24 hours
  Neonatal weight measured after delivery in grams minutes
Apgar score at 1 minute | 1 minute
  Apgar score at 1 minute
Apgar score at 5 minutes | 5 minutes
  Apgar score at 5 minutes
Mode of delivery - questionnaire | up to 24 hours
  Mode of delivery will be recorded as vaginal, assisted (forceps or vacuum), or cesarean

CONTACTS AND LOCATIONS:
Overall Officials: Mrinalini Balki, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No